CLINICAL TRIAL: NCT05744037
Title: Prospective, Multicenter, Open, One-arm Clinical Study of the Safety and Efficacy of the R/R B-NHL Regimen With BTK Inhibitor+Anti-CD19 CAR-T Cells
Brief Title: Clinical Study of the Safety and Efficacy of the R/R B-NHL Regimen With BTK Inhibitor+Anti-CD19 CAR-T Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL365-02
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: B-cell Non Hodgkin Lymphoma
Keywords: BTK inhibitor; Anti CD19 CAR-T cells
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Cell Infusion (Experimental): After FC regimen (fludarabine (25mg/m2/d) on days -5 to -3 and cyclophosphamide (750mg/m2) on days -5) were pretreated, Anti-CD19 CAR T cells were transfused on day 0. The dose was determined by the investigator according to the subjects' own disease conditions and in vitro preparation. Intravenous drip/push at a constant rate for 30 minutes; Ibrutinib, a BTK inhibitor, was enrolled with a standard dose of 560mg qd.
  Interventions: Biological: regimen with BTK inhibitor +Anti-CD19 CAR T cells

INTERVENTIONS:
Biological: regimen with BTK inhibitor +Anti-CD19 CAR T cells — After FC regimen (fludarabine (25mg/m2/d) on days -5 to -3 and cyclophosphamide (750mg/m2) on days -5) were pretreated, Anti-CD19 CAR T cells were transfused on day 0. The dose was determined by the investigator according to the subjects' own disease conditions and in vitro preparation. Intravenous drip/push at a constant rate for 30 minutes; Ibrutinib, a BTK inhibitor, was enrolled with a standard dose of 560mg qd.

SUMMARY:
To evaluate the ORR (CR+PR) of R/R B-NHL subjects treated with BTKi+Anti-CD19 CAR T cells.

DETAILED DESCRIPTION:
The most successful application of CAR-T cell technology in clinical practice is for the treatment of hematologic malignancies, which may be related to the strong specificity of tumor-associated antigen and the weak immunosuppressive effect of tumor microenvironment. CD19 is specifically expressed in B cells and is expressed in all stages of B-cell development and differentiation and in most B-cell tumors, but not in hematopoietic stem cells and other cells. CD19 is a promising target for B-cell tumors and is currently a hot spot in CAR studies.

Antigen-dependent BCR signaling is involved in several downstream pathways, including NF-kB pathway and PI3K/AKT/mTOR pathway, which can promote B cell survival. BTK inhibitors can jointly inhibit the survival of tumor cells by promoting apoptosis and inhibiting the proliferation of tumor cells, reducing the adhesion of tumor cells, and inhibiting chemokines to prevent the migration of B cells.

In this study, BTKi (Ibrutinib) combined with Anti-CD19 CAR-T cells were proposed to treat RR B-NHL, with the main purpose of observing the efficacy and safety of this regimen in patients with relapsed and refractory B-NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the informed consent;
2. Male or female patients aged 18-70 years old;
3. CD19+ B-NHL was confirmed by pathology and histology, and the patient had no effective treatment options at present, such as chemotherapy or hematopoietic stem cell transplantation after recurrence; Or patients voluntarily chose BTKi+Anti-CD19 CAR T as salvage therapy;
4. Subjects showed residual lesions after major treatment and were not suitable for HSCT; Relapse occurs after CR and is not suitable for HSCT; Patients with high risk factors; Relapse or no remission after hematopoietic stem cell transplantation or cellular immunotherapy;
5. Have measurable or evaluable lesions;
6. The patient's main tissues and organs function well;
7. The patient's peripheral shallow venous blood flow is smooth, which can meet the needs of intravenous drip.
8. Patients with ECOG score ≤2, estimated survival time ≥3 months, age ≥ 12 years, ≤ 75 years.

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test is positive) or breastfeeding;
2. Men or women who have planned to get pregnant within the last 1 year;
3. The patients were not guaranteed to take effective contraceptive measures (condom or contraceptive, etc.) within 1 year after enrollment;
4. Patients had uncontrollable infectious diseases within 4 weeks prior to enrollment;
5. Active hepatitis B/C virus;
6. HIV-infected patients;
7. Suffering from a serious autoimmune disease or immunodeficiency disease;
8. The patient is allergic to antibodies, cytokines and other macromolecular biological drugs;
9. The patient had participated in other clinical trials within 6 weeks prior to enrollment;
10. Systemic use of hormones within 4 weeks prior to enrollment (except for inhaled hormones);
11. Suffering from mental illness;
12. The patient has substance abuse/addiction;
13. According to the researchers' judgment, the patient had other conditions that were not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | From 1 month to 1 year.
  CR+PR

SECONDARY OUTCOMES:
Percentage of complete response | From 1 month to 1 year.
  Percentage of complete response
Progression-free survival | From 1 month to 1 year.
  The time between treatment and observation of disease progression or death from any cause.
Duration of response | From 1 month to 1 year.
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No